CLINICAL TRIAL: NCT00079638
Title: Comparative Efficacy Evaluation of Lipid Levels When Treated With Niaspan and Statin or Other Lipid-Modifying Therapies
Brief Title: Comparative Efficacy Evaluation of Lipids When Treated With Niaspan & Statin or Other Lipid-Modifying Therapies-COMPELL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kos Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001-09-03-CR; COMPELL
Record Dates: First submitted 2004-03-10; First posted 2004-03-12 (Estimated); Last update posted 2006-11-01 (Estimated); Status verified 2006-10

CONDITIONS: Dyslipidemia; Coronary Heart Disease; Atherosclerosis; Stroke; Diabetes
Keywords: Niaspan; Niacin; Statin; Cholesterol; Triglycerides; Lipid-Modifying Therapies; Dyslipidemia; Coronary Heart Disease; Atherosclerosis; Stroke; VA-HIT; Niacin Statin Combination Threrapy; High Density Lipoprotein; Low Density Lipoprotein; Hypertension; Diabetes; Adult Treatment Panel III
MeSH Terms: conditions — Dyslipidemias; Coronary Disease; Atherosclerosis; Stroke; Diabetes Mellitus; Hypertension | interventions — Niacin; Atorvastatin; Simvastatin; Ezetimibe; Rosuvastatin Calcium

INTERVENTIONS:
Drug: Niacin
Drug: Atorvastatin
Drug: Simvastatin
Drug: Ezetimibe
Drug: Rosuvastatin

SUMMARY:
The purpose of this study is to evaluate the effectiveness of first-line treatment using Niaspan (an extended release version of niacin) and statins versus other drugs that lower lipid levels, in subjects with elevated fat levels in their blood (dyslipidemia). Statins are a class of medication that is often prescribed to patients who need to lower their cholesterol levels.

DETAILED DESCRIPTION:
Name of Drugs: Niaspan (niacin extended-release tablets), Lipitor® (atorvastatin), Zocor® (simvastatin), Zetia™ (ezetimibe), and Crestor® (rosuvastatin)

Study Treatment: Four open-label parallel treatment groups for 12 weeks of observation

* Niaspan and atorvastatin combination treatment titrated to 2000 mg and 40 mg, respectively;
* combination treatment of simvastatin titrated to 40 mg and ezetimibe maintained at 10 mg;
* rosuvastatin monotherapy treatment titrated to 40 mg; and
* Niaspan and rosuvastatin combination treatment titrated to 1000 mg and 20 mg, respectively.

Objective: To evaluate the relative efficacy of first-line therapy using the combination of Niaspan and atorvastatin versus the combination of simvastatin and ezetimibe versus rosuvastatin monotherapy versus the combination of Niaspan and rosuvastatin in patients with dyslipidemia.

Population:

* Male or female patients 21 years of age or older
* Patients who are eligible for treatment based upon National Cholesterol Education Program Adult Treatment Panel III (NCEP-ATP III) recommendations at the end of the Qualification period;
* All patients must have mean triglycerides (TG) ≤ 300 mg/dL.

Design: A Phase IV, 12-week, randomized, multi-center, open-label, four-arm, parallel-group study evaluating the efficacy of Niaspan and statin therapy versus other lipid-modifying therapies preceded by a four-week washout of any previous lipid-lowering therapy.

ELIGIBILITY:
Inclusion Criteria:

All of the following criteria must be answered "Yes":

1. Patient is 21 years of age or older and willing to participate for the duration of the study;
2. Patient has read, signed, and agreed to the items listed in the informed consent form and HIPAA authorization form prior to the initiation of any study procedures and/or discontinuing any medications;
3. Patient is eligible for treatment following the drug washout period based upon the NCEP ATP III entry criteria and the LDL-C variability ≤ 15%;
4. Patient has mean triglyceride level (TG) ≤ 300 mg/dL;
5. Patient is willing to withdraw from any current anti-dyslipidemic medications or other prohibited medication for approximately 6 weeks prior to randomization (4 weeks prior to qualification visits) and for the duration of the study;
6. If the patient is female, the patient must not be pregnant or breast-feeding and not planning to become pregnant or to breast-feed for the duration of the study. Women of childbearing potential must commit to using a medically acceptable method of birth control such as oral contraception, intrauterine device (IUD), or a double-barrier method of contraception. Women using oral contraception must have done so for at least 3 months prior to randomization, and continue to do so for the duration of the study. To be considered not of childbearing potential, women must be post-menopausal for at least 2 years or surgically sterile.

Exclusion Criteria:

All the following criteria must be answered "No":

1. Patient has an allergy, hypersensitivity, or intolerance to niacin, simvastatin, atorvastatin, ezetimibe, rosuvastatin or their derivatives;
2. Patient drinks more than 14 alcoholic drinks per week or has a previous history (within 12 months of screening) of substance abuse or dependency;
3. Patient has untreated or unsuccessfully treated psychiatric disease;
4. Patient has used an investigational study medication or participated in an investigational study within 30 days of obtaining qualification labs;
5. Patient has taken a prohibited medication within 4 weeks of obtaining qualification labs for the study (See section 8.0 - Concomitant Medications);
6. Patient has a history of any of the following:

   * active gallbladder disease within the preceding 12 months (cholecystectomy is allowed);
   * pancreatitis;
   * liver disease (e.g., hepatitis B and/or C);
   * persistent uncontrolled or untreated severe hypertension;
   * Type I or Type II diabetes;
   * persistent uncontrolled or untreated hypothyroidism;
   * arterial bleeding;
   * unstable angina;
   * myocardial infarction, coronary artery bypass graft surgery, or angioplasty within the preceding 6 months;
   * stroke, transient ischemic attack (TIA), or deep vein thrombosis (DVT) within the preceding 6 months;
   * congestive heart failure NYHA class III or IV;
   * active cancer within the last 5 years or a diagnosis of cancer within the last 5 years (excluding basal cell carcinoma);
   * fibromyalgia, myopathy, rhabdomyolysis, unexplained muscle pain or weakness, and/or discontinuation of a statin because of myalgia; and/or
   * life expectancy < 2 years.
7. Patient has any of the following abnormalities at any of the Screening or Qualification Visits:

   * CPK elevation > 3xULN;
   * aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 1.3xULN;
   * serum creatinine ≥ 1.5 mg/dL;
   * creatinine clearance < 30 mL/min, as calculated using the Cockroft and Gault formula by the central laboratory;
   * active gout symptoms and/or uric acid level > 1.3xULN;
   * and/or active peptic ulcer disease;
8. Patient is planning to undergo major surgery within the next 6 months;
9. Patient has any health condition or laboratory abnormality that, in the opinion of the Principal Investigator, may be adversely affected by the procedures or medications in this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-04; Study Completion 2005-05

PRIMARY OUTCOMES:
Mean percent change in LDL-C from Baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: COMPELL TEAM, Principal Investigator — Contact COMPELL Team Member (800) 722-4567